CLINICAL TRIAL: NCT01197235
Title: Prevention of Contrast-Induced Nephropathy by Darbepoetin in Patients With Chronic Kidney Disease
Brief Title: Effect of Darbepoetin in Contrast-induced Nephropathy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: difficult to enroll targeted participants
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Ki Young Na, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SNUBH B- 0811/063-001
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Acute Kidney Injury
Keywords: darbepoetin, chronic kidney disease, coronary angiography
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- darbepoetin-α (Experimental): Infusion of darbepoetin-α 1.5 μg/kg will be performed 1 hour before angiography
  Interventions: Drug: darbepoetin-α
- isotonic saline (Placebo Comparator): Infusion of isotonic saline will be performed 1 hour before angiography
  Interventions: Drug: isotonic saline

INTERVENTIONS:
Drug: darbepoetin-α — Infusion of darbepoetin-α 1.5 μg/kg will be performed 1 hour before angiography
  Other Names: aranesp
  Arms: darbepoetin-α
Drug: isotonic saline — Infusion of isotonic saline will be performed 1 hour before angiography
  Other Names: 0.9% NaCl solution
  Arms: isotonic saline

SUMMARY:
The purpose of this study is to determine whether the drug that produce red blood cells is effective in the prevention of kidney dysfunction after coronary angiography in patients with chronic kidney disease.

DETAILED DESCRIPTION:
Use of radiocontrast agent is inevitable in computed tomography or angiography. However, contrast agent can aggravate kidney function. Contrast-induced nephropathy (CIN) refers to the clinical situation where decreased kidney function after use of contrast. CIN is the 3rd most common cause of acute kidney injury in the hospitals. There are a lot of reports that death rate is increased in patients with CIN.

Erythropoietin is an agent that treat anemia. It also has been reported to have a tissue-protective effect in the animal experiments.

In this study, we hypothesized that erythropoietin can reduce the incidence of CIN in patients with chronic kidney disease undergoing coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 yr
* estimated glomerular filtration rate (GFR) < 60 ml/min/1.73m2

Exclusion Criteria:

* Chronic renal replacement therapy (hemodialysis, peritoneal dialysis, continuous renal replacement therapy)
* Pregnancy or lactation
* Use of contrast agent within 1 week
* Emergent CAG or PCI
* Not recovered from AKI(acute kidney injury)
* Use of nephrotoxic drugs within 48 hr
* Cardiogenic shock (SBP(systolic blood pressure) < 90 mmHg) or pulmonary edema
* Uncontrolled hypertension (SBP ≥ 200 mmHg or DBP(diastolic blood pressure) ≥ 130 mmHg)
* History of hypersensitivity to contrast agent
* Known allergy or hypersensitivity to EPO(erythropoietin)
* Use of EPO within 1 month
* Anemia (hemoglobin < 9 g/dL)
* Ventilatory care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
incidence of contrast-induced nephropathy (CIN) | 48 hours
  a greater than 25 percent increase in serum Cr or an absolute increase in serum Cr of 0.5 mg/dL within 48 hours after using the contrast agent

SECONDARY OUTCOMES:
maximum difference in Cr levels before and after CAG(coronary angiography) or PCI(percutaneous coronary intervention) | 1 month after the intervention
  the maximum difference in Cr levels before and after CAG or PCI, the incidence of AKI requiring renal replacement therapy, length of hospital stay, mortality, myocardial infarction, revascularization, and the occurrence of stroke

CONTACTS AND LOCATIONS:
Overall Officials: Ki Young Na, MD PhD, Principal Investigator — Seoul Ntional University Bundang Hospital, Seoul National University College of Medicine
Locations (1):
- Seoul National University Bundang Hospital,, Seongnam, South Korea